CLINICAL TRIAL: NCT05954169
Title: A Single-dose, Open-label/Pharmacokinetic and Safety Study of SHR4640 in Subjects With Moderate Renal Insufficiency and Healthy Subjects
Brief Title: Pharmacokinetic/Pharmacokinetic and Safety Studies of SHR4640 in Subjects With Moderate Renal Insufficiency and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR4640-111
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — ruzinurad

STUDY DESIGN:
Intervention Model Description: Single-dose, open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A in moderately renal insufficiency subjects (Experimental)
  Interventions: Drug: SHR4640
- Treatment group B in healthy subjects (Experimental)
  Interventions: Drug: SHR4640

INTERVENTIONS:
Drug: SHR4640 — SHR4640 single-dose

SUMMARY:
This study aimed to evaluate the pharmacokinetics, pharmacodynamics, and safety of SHR4640 tablets in subjects with moderate renal insufficiency and healthy subjects, and to explore the relationship between renal function (e.g., eGFR) and SHR4640 pharmacokinetic and pharmacodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

-

Moderate renal impaired subjects:

1. Able and willing to provide a written informed consent.
2. 18 years to 65 years (inclusive).
3. Body mass index should be between 18 and 35 kg/m2 (inclusive).
4. eGFR should be between 30 and 59 mL/min/1.73 m2 (inclusive).
5. The renal function status is stable, and the results of two eGFR tests during the screening period (at least 3 days apart, but within 14 days) should be within ±25%.
6. If subjects with underlying diseases required drug treatment, the dose needs to be kept stable during study.

Healthy subjects:

1. Able and willing to provide a written informed consent.
2. 18 years to 65 years (inclusive).
3. Body mass index should be between 18 and 35 kg/m2 (inclusive).
4. eGFR should be ≥ 90 and < 130 mL/min/1.73 m2.
5. The renal function status is stable, and the results of two eGFR tests during the screening period (at least 3 days apart, but within 14 days) should be within ±25%.

Exclusion Criteria:

-

Moderate renal impaired subjects:

1. Pregnant or nursing women.
2. No birth control 2 weeks before screening or until one week after SHR4640 administration.
3. Average daily alcohol consume more than 14g for female or more than 28g for male within 1 month before screening, or baseline alcohol screening is positive.
4. Smokers (average daily smoking of 10 cigarettes or more in the 3 months before screening).
5. Subject with a history of substance abuse and drug abuse.
6. The investigators determined that other conditions were inappropriate for participation in this clinical trial.
7. The investigators or relevant staff of the research centers or others directly involved in the study.
8. 2 weeks before SHR4640 administration sUA level ≥480 μmol/L.
9. Alanine aminotransferase and/or aspartate aminotransferase>2×ULN, alkaline phosphatase (ALP)>2.5×ULN.
10. Positive result for hepatitis B surface antigen.
11. Positive result for human immunodeficiency virus (HIV), hepatitis C virus antibody or syphilis antibody.
12. White blood cell < 3.0×109/L, and/or hemoglobin <80 g/L, and/or platelet <80×109/L.
13. 12-lead electrocardiogram (ECG) showed abnormal and clinically significant.
14. History of hypersensitivity to SHR4640 or its analogues.
15. History or suspected crystals or stones in the urinary system during the screening period of B-ultrasound.
16. History of been diagnosed with acute kidney injury in the past or screening period.
17. History of kidney transplantation.
18. Renal dialysis required during the study.
19. Urinary incontinence or anuria (eg< 100 mL/d).
20. Cardiovascular, neuropsychiatric, respiratory, digestive tract, endocrine and other systemic diseases within 1 year before screening, which were judged to be serious by the investigators.
21. Have grade III or IV congestive heart failure (New York Heart Association classification) or myocardial infarction, unstable angina, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage or transient ischemic attack within 1 year of screening, and other cardiovascular and cerebrovascular events leading to hospitalization.
22. History of active peptic ulcer within 1 year before screening, previous history of active gastrointestinal bleeding, gastrointestinal perforation, history of inflammatory bowel disease, or active peptic ulcer at screening.
23. Have a malignant tumor, or have a history of malignant tumor within 5 years before screening.
24. SBP≥180 mmHg and/or DBP ≥110 mmHg.
25. Had undergone major surgery within 3 months prior to screening, or have not recovered from surgery, or plan major surgery during the study.
26. Received the last dose of a study drug (or treatment with a medical device) within 3 months or 5 T1/2 (whichever is longer) of the screening or are currently participating in another study of a study drug (or medical device).
27. Blood donation within 1 month before screening; Or patients with trauma or major surgical procedures who donated blood or lost blood ≥400 mL in the 3 months prior to screening.
28. Has unsuitable venous for blood sampling.
29. Use of any of the following, unless agreed as nonclinically relevant by the Investigator and the Sponsor:

1) Use of any over the-counter, nutraceuticals, or prescription medications that might interfere with the absorption, distribution, metabolism, or excretion of SHR4640 (proton-pump inhibitor, fluconazole, indomethacin, ranitidine, flurbiprofen, probenecid, aprepitant, etc.) within 2 weeks of screening.

2) Unstable dosage of urate-lowering drugs within 6 weeks of Day 1. 3) Diuretics within 2 weeks of Day 1. 4) Aspirin in excess of 100 mg daily or unstable dose within the 2 weeks of Day 1.

5) Unstable dosage of antihypertensive, lipid-lowering and hypoglycemic drugs within 2 weeks of Day 1.

6) Have received or been exposed to other live vaccines or live attenuated vaccines within 3 months prior to Day 1, or who plan to receive live vaccines or live attenuated vaccines during the study.

30. Consumes grapefruit and/or poppy seed within 48 hours before SHR4640 administration.

31. Taken prescription drugs, over-the-counter drugs, herbal medicines or food supplements other than drugs for the treatment of renal insufficiency and other concomitant diseases within 2 weeks before Day 1.

Healthy subjects:

1. Pregnant or nursing women.
2. No birth control 2 weeks before screening or until one week after SHR4640 administration.
3. Average daily alcohol consume more than 14g for female or more than 28g for male within 1 month before screening, or baseline alcohol screening is positive.
4. Smokers (average daily smoking of 10 cigarettes or more in the 3 months before screening).
5. Subject with a history of substance abuse and drug abuse.
6. The investigators determined that other conditions were inappropriate for participation in this clinical trial.
7. The investigators or relevant staff of the research centers or others directly involved in the study.
8. 2 weeks before SHR4640 administration sUA level ≥420 μmol/L.
9. Laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function) during the screening period were abnormal and the investigators determined that they were clinically significant.
10. Positive result for hepatitis B surface antigen.
11. Positive result for human immunodeficiency virus (HIV), hepatitis C virus antibody or syphilis antibody.
12. 12-lead electrocardiogram (ECG) showed abnormal and clinically significant.
13. History of hypersensitivity to SHR4640 or its analogues.
14. History or suspected crystals or stones in the urinary system during the screening period of B-ultrasound.
15. History of been diagnosed with chronic or acute kidney injury in the past or screening period. History of kidney transplantation.
16. Cardiovascular, neuropsychiatric, respiratory, digestive tract, endocrine and other systemic diseases within 1 year before screening, which were judged to be serious by the investigators.
17. Have a malignant tumor, or have a history of malignant tumor within 5 years before screening.
18. SBP>140 mmHg or <90 mmHg and/or DBP >90 mmHg or <60 mmHg.
19. Had undergone major surgery within 3 months prior to screening, or have not recovered from surgery, or plan major surgery during the study.
20. Received the last dose of a study drug (or treatment with a medical device) within 3 months or 5 T1/2 (whichever is longer) of the screening or are currently participating in another study of a study drug (or medical device).
21. Blood donation within 1 month before screening; Or patients with trauma or major surgical procedures who donated blood or lost blood ≥400 mL in the 3 months prior to screening.
22. Has unsuitable venous for blood sampling.
23. Use of any of the following, unless agreed as nonclinically relevant by the Investigator and the Sponsor:

1) Use of any over the-counter, nutraceuticals, or prescription medications that might interfere with the absorption, distribution, metabolism, or excretion of SHR4640 (proton-pump inhibitor, fluconazole, indomethacin, ranitidine, flurbiprofen, probenecid, aprepitant, etc.) within 2 weeks of screening.

2) Use of urate-lowering drugs within 6 weeks of Day 1. 3) Have received or been exposed to other live vaccines or live attenuated vaccines within 3 months prior to Day 1, or who plan to receive live vaccines or live attenuated vaccines during the study.

24. Consumes grapefruit and/or poppy seed within 48 hours before SHR4640 administration.

25. Taken any prescription drugs, over-the-counter drugs, herbal medicines or food supplements within 2 weeks before Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
PK parameters of SHR4640: Cmax | 0 hour to 72 hour after administration
PK parameters of SHR4640: AUC0-t | 0 hour to 72 hour after administration
PK parameters of SHR4640: AUC0-inf | 0 hour to 72 hour after administration

SECONDARY OUTCOMES:
PK parameters of SHR4640: Tmax | 0 hour to 72 hour after administration
PK parameters of SHR4640: t1/2 | 0 hour to 72 hour after administration
PK parameters of SHR4640: CL/F | 0 hour to 72 hour after administration
PK parameters of SHR4640: Vz/F | 0 hour to 72 hour after administration
Amount of SHR4640 excreted in urine (Ae0-72h) | 0 hour to 72 hour after administration
Serum uric acid concentration | 0 hour to 72 hour after administration
Amount of uric acid excreted in urine | 0 hour to 72 hour after administration
Adverse events | from ICF signing date to approximate day 8

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided